CLINICAL TRIAL: NCT05355285
Title: Type 1 Diabetes and Depression: Role of Brain Glutamate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas Bolo, Director of Neuroimaging in Psychiatry, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NIH R01-DK084202
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Type1diabetes; Depressive Symptoms; Major Depressive Disorder
Keywords: Hyperglycemia; Euglycemic hyperinsulinemic clamp; Euglycemia; Magnetic Resonance Spectroscopy; Magnetic Resonance Imaging; Glutamate
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Hyperglycemia | interventions — Glucose Clamp Technique

STUDY DESIGN:
Intervention Model Description: There are 4 subject groups for this study: 1) T1DM without current depressive symptoms with no history of major depressive disorder; 2) T1DM with current depressive symptoms and with a history of major depressive disorder; 3) Non-diabetic controls without current depressive symptoms and with no history of major depression; 4) Non-diabetic controls with current depressive symptoms and with major depression history. For all subjects, MRS brain glutamate is assessed during basal euglycemia, and for a subset of subjects per group, during an acute hyperglycemic clamp. To control for potential confounding effects of hyperinsulinemia, brain glutamate is also assessed during a euglycemic hyperinsulinemic clamp in a subset of controls (group 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Euglycemia (Experimental): Subjects with T1DM (Groups 1 and 2): 1) receive a low dose insulin infusion to reduce their plasma glucose to euglycemia; 2) receive a continuous infusion of insulin at the rate of 0.25 milli-Units/kg/min to maintain euglycemia during a Baseline MRI scanning period.
  Subjects without diabetes (Groups 3 and 4) are scanned during a Baseline MRI scanning period (no intervention is needed to maintain euglycemia in these subjects).
  Interventions: Procedure: Glucose Clamp
- Hyperglycemic Clamp (Experimental): Subjects with T1DM (Groups 1 and 2): 1) receive a primed variable glucose infusion to attain a target increase in glycemic level of +5.5 mmol/L; 2) receive a continuous infusion of insulin at the rate of 0.25 milli-Units/kg/min.
  Subjects without diabetes (Groups 3 and 4): 1) receive a primed variable glucose infusion to attain a target increase in glycemic level of +5.5 mmol/L.
  Interventions: Procedure: Glucose Clamp
- Hyperinsulinemic Euglycemic Clamp (Experimental): Subjects without diabetes or depression (Group 3) have a second study visit at least 15 days after the Hyperglycemic Clamp visit. They receive a variable insulin infusion to match individual insulin levels to the levels attained during the Hyperglycemic Clamp and they receive a variable glucose infusion to maintain euglycemia.
  Interventions: Procedure: Glucose Clamp

INTERVENTIONS:
Procedure: Glucose Clamp — Subjects receive variable rates of glucose or insulin infusions to adjust and maintain desired plasma glucose or insulin levels.
  Other Names: Hyperglycemic, Euglycemic, or Hyperinsulinemic Euglycemic Clamp

SUMMARY:
The goal of this study is to examine the effect of chronic and acute hyperglycemia in type 1 diabetes mellitus (T1DM) on brain glutamate levels using magnetic resonance spectroscopy (MRS), and associations of brain glutamate with symptoms of depression.

DETAILED DESCRIPTION:
The research of this study is focused on elucidating the relationship between the perturbations in glucose metabolism associated with T1DM and the higher prevalence of major depressive episodes in this patient population. Converging evidence associating high brain levels of glutamate with T1DM and depression leads to the hypothesis that the link between diabetes-related glucose metabolic disorders and depression is excessive brain glutamate. The overarching aim of the study is to examine the effect of chronic and acute hyperglycemia in T1DM on brain glutamate levels. Four subject groups were studied and characterized: T1DM patients with and without concurrent depressive symptoms, and non-diabetic subjects with and without concurrent depressive symptoms. Two brain regions were examined : the anterior cingulate cortex (ACC), known to play an essential role in the regulation of emotions, and a control occipital cortex region. Regional brain glutamate concentrations were measured using high-field (3 Tesla) localized multidimensional magnetic resonance spectroscopy (MRS), regional indices of brain function were assessed using functional magnetic resonance imaging (fMRI), concurrent depression symptom severity and depression history were evaluated using psychiatric assessment, extensive medical evaluation of patients was performed including evaluation of glycemic control (HbA1c), evaluation of behavioral performance on emotional and cognitive tasks and evaluation of regional brain cortical thickness using high-resolution structural MRI. For all subjects, MRS brain glutamate was assessed during basal euglycemia and, for a subset of subjects per group, during an acute hyperglycemic clamp. To control for potential confounding effects of hyperinsulinemia, brain glutamate was also assessed during a euglycemic hyperinsulinemic clamp in a subset of healthy controls without diabetes or depressive symptoms.

ELIGIBILITY:
T1DM Subjects:

Inclusion Criteria:

* 10-25 years duration of T1DM.
* Relatively low levels of complications from diabetes.

Exclusion Criteria:

* Type 2 diabetes and/or gestational diabetes.
* Other major clinical conditions such as cancer, symptomatic coronary artery disease, (e.g., prior myocardial infarction), stroke, proliferative diabetic retinopathy requiring a laser treatment, clinically significant diabetic nephropathy as evidenced by urinary albumin levels > 300 mg/day and/or serum creatinine > 1.5 mg/dl for men and > 1.4 mg/dl for women, painful or symptomatic neuropathy, and/or diagnosed gastroparesis.
* Current or past history of attention deficit hyperactivity disorder, bipolar disorder, obsessive compulsive disorder, panic disorder, substance dependence or schizophrenia.
* Ethanol dependence and/or nicotine dependence according to Diagnostic and Statistical Manual-IV criteria and heavy smokers according to the Epidemiology of Diabetes Interventions and Complications scale 57.

Control Subjects:

Inclusion Criteria:

* No history of T1DM or Major Depressive Disorder.
* Normal fasting blood glucose, HbA1c and hematocrit levels.

Exclusion Criteria:

* Known chronic medical illness such as rheumatoid arthritis or major cardiac, kidney or liver disease or anemia.
* Current or past history of attention deficit hyperactivity disorder, bipolar disorder, obsessive compulsive disorder, panic disorder, substance dependence or schizophrenia.
* Past history of a major depressive episode, as well as with current symptoms of depression as defined by a HAMD-17 score ≥ 10.

Subjects with depressive history and current depressive symptoms:

Inclusion criteria:

* History of at least one episode of major depression.
* A 17-item HAM-D (HAMD-17) score ≥ 10 and ≤ 27

Exclusion criteria:

* Current or past history of attention deficit hyperactivity disorder, bipolar disorder, obsessive compulsive disorder, panic disorder, substance dependence or schizophrenia.
* Subjects under current treatment with antidepressant medication.
* Subjects with acute severe depression or acute suicidal ideation, who in the opinion of the psychiatrist are clinically inappropriate for participation in the study.
* Subjects who in the opinion of the psychiatrist are clinically inappropriate for a one-week delay in antidepressant medication treatment.
* HAMD-17 score > 27.

All Subjects:

Exclusion criteria related to MR procedure:

Participants who have metal in their body, suffer from claustrophobia or panic disorder or women who are pregnant, or who are currently breast-feeding cannot participate in this research study.

Additional MR exclusion criteria include people with:

* Cardiac pacemakers
* Metal clips on blood vessels (also called stents)
* Artificial heart valves
* Artificial arms, hands, legs, etc.
* Brain stimulator devices
* Implanted drug pumps
* Ear implants
* Eye implants or known metal fragments in eyes
* Exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others)
* Other metallic surgical hardware in vital areas
* Certain tattoos with metallic ink (subjects are requested to inform the investigator if they have a tattoo)
* Certain transdermal (skin) patches such as NicoDerm (nicotine for tobacco dependence), Transderm Scop (scopolamine for motion sickness), or Ortho Evra (birth control).
* Claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Anterior cingulate cortex glutamate concentration during Baseline Euglycemia | Baseline Euglycemia
  mmol/kg wet weight of brain tissue
Change in anterior cingulate cortex glutamate concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue

SECONDARY OUTCOMES:
Change in anterior cingulate cortex glutamate concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in occipital lobe glutamate concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in occipital lobe glutamate concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in anterior cingulate cortex myo-inositol concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in anterior cingulate cortex myo-inositol concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in occipital lobe myo-inositol concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in occipital lobe myo-inositol concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  mmol/kg wet weight of brain tissue
Change in Intrinsic Neuronal Activity from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  Fractional amplitude of low frequency fluctuations (fALFF) of fMRI signal
Change in Intrinsic Neuronal Activity from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  Fractional amplitude of low frequency fluctuations (fALFF) of fMRI signal
Change in Functional Connectivity from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  Correlation strength of fMRI signal fluctuations between brain regions
Change in Functional Connectivity from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  Correlation strength of fMRI signal fluctuations between brain regions
Change in plasma glucose concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  mmol/L
Change in plasma glucose concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  mmol/L
Change in plasma insulin concentration from Baseline Euglycemia to Hyperglycemia | During the MRI scanning visit with hyperglycemic clamp, up to 180 minutes
  micro-Unit/mL
Change in plasma insulin concentration from Baseline Euglycemia to Hyperinsulinemic Euglycemia | During the MRI scanning visit with hyperinsulinemic euglycemic clamp, up to 180 minutes
  micro-Unit/mL

OTHER OUTCOMES:
Hamilton Depression rating (HAM-D) | Baseline
  Hamilton depression rating Score from 0 to 51. Higher scores indicate worse depression.
Revised Symptom Checklist rating (SCL-90-R) | Baseline
  Revised Symptom Checklist rating Score from 0 to 360. Higher scores indicate worse symptoms.
Wechsler Abbreviated Scale of Intelligence - intelligence quotient (WASI-IQ) | Baseline
  Wechsler Abbreviated Scale of Intelligence - intelligence quotient Score from 40 to 160 (mean = 100, standard deviation = 15). Higher scores indicate better intellectual ability.
Grooved Pegboard task time | Baseline
  seconds
HbA1c | Baseline
  Percentage
BMI | Baseline
  kg/m2
Emotional Stroop Task response time | Baseline
  milli-seconds
Self Referential Emotional Task (SRET) response time | Baseline
  milli-seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas R Bolo, PhD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bolo NR, Jacobson AM, Musen G, Keshavan MS, Simonson DC. Acute Hyperglycemia Increases Brain Pregenual Anterior Cingulate Cortex Glutamate Concentrations in Type 1 Diabetes. Diabetes. 2020 Jul;69(7):1528-1539. doi: 10.2337/db19-0936. Epub 2020 Apr 15. PMID 32295804
- [Result] Bolo NR, Jacobson AM, Musen G, Simonson DC. Hyperglycemia and hyperinsulinemia effects on anterior cingulate cortex myoinositol-relation to brain network functional connectivity in healthy adults. J Neurophysiol. 2022 May 1;127(5):1426-1437. doi: 10.1152/jn.00408.2021. Epub 2022 Apr 13. PMID 35417272